CLINICAL TRIAL: NCT02525666
Title: Evaluation of Bilateral Laparoscopic Repair of Groin Hernias With One Large Self-fixating Mesh (ProGripTM) in a Prospective Cohort Study
Brief Title: Bilateral Laparoscopic Repair of Groin Hernias With One Large Self-fixating Mesh (ProGripTM)
Acronym: BigWig
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Head of the Department of Surgery, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: BigWig Study
Record Dates: First submitted 2015-08-05; First posted 2015-08-17 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Hernia; Recurrence; Quality of Life
MeSH Terms: conditions — Hernia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigation of a bilateral inguinal hernia repair using one large self-fixating mesh covering both groins. Health outcomes are assessed using different questionaires with focus on urinary symptoms (with ICIQ-MLUTS score), the recurrence rate, postoperative pain measurement, and Quality of Life assessment with EuraHS-QoL and chronic pain monitoring for 12 months.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Evidence in groin hernia repair showed a significant reduction in recurrence rates since the introduction of mesh repair. Hence all current guidelines state that in surgical treatment of groin hernias in adults a mesh should be used.

   In laparoscopic groin hernia repair a mesh is positioned in the preperitoneal plane. Two techniques are commonly used. A transabdominal technique (TransAbdominal PrePeritoneal - TAPP), in which the preperitoneal plane is dissected throughout the abdomen, with a closure of the peritoneum after positioning of the mesh, and a preperitoneal technique (Totally ExtraPeritoneal - TEP) in which the peritoneum remains intact.

   Fixation of the mesh was originally performed by penetrating fixation, using staples or tackers. Alternative fixation with glue, self-fixating meshes or no mesh fixation at all, have been proposed to avoid the postoperative pain related to the penetrating fixation. Several studies were not able to show significant differences in recurrence rates between the different mesh fixation techniques. In general, sufficient overlap seems more important than fixation of the mesh. However, current guidelines state that tacker or suture fixation of the mesh for groin hernia should be avoided.

   Concerns are often raised about large medial hernias (EHS classification: M3) because the medial overlap of the mesh beyond the hernia defect is small. An overlap of less than 2-3 cm may lead to protrusion of the mesh in the hernia opening, and this risk is increased in large direct hernias. In general, the larger the hernia opening, the more overlapping there should be. Observational studies have shown a higher recurrence rate in the repair of direct (i.e. medial) hernias. In a recent consensus statement, Poelman et al. stated that diverse types of inguinal hernias (direct vs. indirect, large vs. small) should be distinguished and treated in a different way. Despite the fact that randomized trials did not differentiate between large or small hernias, they state that the use of a heavy weight mesh, mesh fixation or larger mesh size should be considered in case of large medial hernias.

   In repair of bilateral inguinal hernias, current guidelines state that laparoscopic treatment is the preferable approach, without clear advantage of TEP over TAPP or vice-versa. During transabdominal (TAPP) repair, evaluation and subsequent treatment of a contralateral hernia can be performed without additional incision and/or trocar placement. Whether one large mesh or two separate meshes with sufficient overlap should be used, remains unclear. The IEHS guidelines state that both options can be used. However, the recurrences detected after the use of two separate meshes suggest the presence of weaker zone at the midline, despite the overlap. On the other hand, application of one large mesh seems to be technically more difficult. In laparoscopic groin hernia repair, the mesh is placed in the anatomical space between pubic bone and bladder. Any type of mesh might therefore potentially influence the urinary bladder function. Until now it is not clear if these urinary symptoms will be different in patients with one large mesh compared to those with two overlapping meshes.
2. AIM AND DESIGN OF THE STUDY Purpose of this study is the assessment urinary symptoms after bilateral repair using one large self-fixating mesh covering both groins in repair of bilateral inguinal hernias. Health outcomes are assessed using different questionaires with focus on urinary symptoms (with ICIQ-MLUTS score), the recurrence rate, postoperative pain measurement, and Quality of Life assessment with EuraHS-QoL and chronic pain monitoring for 12 months.

   A total of 100 male patients will be entered in the trial in AZ MARIA MIDDELARES, for which an inclusion period of 24 months is anticipated. Study inclusion will be based on clinical examination and/or ultrasonography. Informed Consent will be obtained pre-operatively.
3. OPERATIVE STANDARD PROCEDURES A bilateral laparoscopic groin hernia repair will be performed, using one large self-fixating mesh (ProGripTM). in transabdominal (TAPP) approach or in totally extra-peritoneal (TEP) approach on all patients.
4. FOLLOW-UP After receiving informed consent and planned surgery, patients will get invited for a standard clinical check-up (at 1 month en 12 months post-operatively) and for assessment of urinary symptoms using the ICIQ-MLUTS (International Consultation on Incontinence modular Questionnaire on Lower Urinary Tract Symptoms) at 1 month, 3 months en 12 months post-operatively.

   Recurrence rates will be based on clinical examination by the surgeon during follow-up. In case of uncertainty during clinical evaluation further investigation using ultrasonography and/or CT scan will be performed.

   Quality of Life, using the pre- and postoperative EuraHS-QoL score and postoperative pain using a VAS (Visual Analogue Scale) scale will be assessed during the clinical follow-up moments. Additional registration of pain medication used will be performed.
5. DATA COLLECTION AND ANALYSIS All data related to the surgical procedure, patient comorbidities and the post-operative course will be documented prospectively. Anonymized data of all patients will be collected in the online platform EuraHS (European Registry of Abdominal Wall Hernias), developed by the scientific working of European Hernia Society EHS under a specific study account.

A study specific CRF including the ICIQ-MLUTS, the EuraHS-QoL, the VAS (visual analog scale) and VRS (verbal rating scale will be provided by the trial secretariat and gathered by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for primary bilateral inguinal hernia repair

Exclusion Criteria:

* recurrent groin hernia
* open hernia repair
* unilateral hernias
* concomitant repair of another abdominal hernia e.g. umbilical hernia
* hernia repair combined with another surgical procedure
* emergency operations, like incarcerated hernias
* patients under the age of 18 years or over 80 years
* ASA score 4 or more
* patients unable to perform the QoL assessment, because of language barrier or intellectual incapacity
* no informed consent of the patient

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients, men only, ages between 18 and 80 years with a primary bilateral inguinal hernias will be included based on clinical examination and/or ultrasonography.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Assessment of ICIQ-MLUTS Score | 12 months
  Assessment of urinary symptoms with the ICIQ_MLUTS score at 12 month after laparoscopic repair of bilateral inguinal hernia

SECONDARY OUTCOMES:
Assessment of ICIQ-MLUTS Score | preoperative, 1 month and 3 month post-operative
  Assessment of urinary symptoms with the ICIQ_MLUTS score (pre-operatively, 1 and 3 month postoperatively)
Quality of Life assessment | pre-operatively, 1, 3 and 12 month postoperatively
  Quality of Life assessment with the EuraHS QoL score (pre-operatively, 1, 3 and 12 month postoperatively)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

REFERENCES:
- [Background] Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia. 2009 Aug;13(4):343-403. doi: 10.1007/s10029-009-0529-7. Epub 2009 Jul 28. PMID 19636493
- [Background] Poelman MM, van den Heuvel B, Deelder JD, Abis GS, Beudeker N, Bittner RR, Campanelli G, van Dam D, Dwars BJ, Eker HH, Fingerhut A, Khatkov I, Koeckerling F, Kukleta JF, Miserez M, Montgomery A, Munoz Brands RM, Morales Conde S, Muysoms FE, Soltes M, Tromp W, Yavuz Y, Bonjer HJ. EAES Consensus Development Conference on endoscopic repair of groin hernias. Surg Endosc. 2013 Oct;27(10):3505-19. doi: 10.1007/s00464-013-3001-9. Epub 2013 May 25. No abstract available. PMID 23708718
- [Background] Tam KW, Liang HH, Chai CY. Outcomes of staple fixation of mesh versus nonfixation in laparoscopic total extraperitoneal inguinal repair: a meta-analysis of randomized controlled trials. World J Surg. 2010 Dec;34(12):3065-74. doi: 10.1007/s00268-010-0760-5. PMID 20714896
- [Background] Donovan JL, Peters TJ, Abrams P, Brookes ST, de aa Rosette JJ, Schafer W. Scoring the short form ICSmaleSF questionnaire. International Continence Society. J Urol. 2000 Dec;164(6):1948-55. PMID 11061889
- [Derived] Muysoms F, Dewulf M, Kyle-Leinhase I, Baumgartner R, Ameye F, Defoort B, Pletinckx P. Laparoscopic bilateral groin hernia repair with one large self-fixating mesh: prospective observational study with patient-reported outcome of urological symptoms and EuraHS-QoL scores. Surg Endosc. 2020 Feb;34(2):920-929. doi: 10.1007/s00464-019-06850-7. Epub 2019 May 28. PMID 31139996